CLINICAL TRIAL: NCT01749046
Title: Double-blind, Placebo-controlled Clinical Study to Evaluate the Efficacy, Safety and Tolerability of a Fixed Dose of Remegal as Adjunctive Therapy in Patients With Partial Seizures
Brief Title: Remegal Fixed Dose as Adjunctive Therapy in Patients With Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valexfarm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-MPP02EPI; 11-МРР02ЕРI (Other: Ministry of Health of Russian Federation)
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Epilepsy; Simple Partial Seizures; Complex Partial Seizures; Partial Seizures With Secondary Generalization
Keywords: Epileptic seizures, Partial seizures
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Seizures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remegal (Experimental): Remegal 1500 mg
  Interventions: Drug: Remegal
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Remegal

INTERVENTIONS:
Drug: Remegal — Remegal 1500 mg for 12 weeks
  Other Names: Beprodon; AED

SUMMARY:
The purpose of this study is to determine weather Remegal in fixed dosage 1500 mg/daily is effictive and safe in patients with epilepsy with partial seizures

DETAILED DESCRIPTION:
Phase III

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, aged from 18 to 65
* Diagnosis of epilepsy with simple and/or complex partial seizures both with or without secondary generalization based on the ILAE classification
* Results of at least one prior electroencephalogram (EEG) and magnetic resonance imaging (MRI)/computerized tomography scan no more than 5 years should confirm the diagnostic of partial seizures
* If seizures are simple partial ones, only patients with motor signs must be enrolled
* The onset date of partial seizures according to patient's report must be at least 2 years
* The patient must report an average of at least 8 partial seizures per 56 days prior to the baseline visit
* The patient must not have seizure-free period longer than 21 days during the 8 weeks prior to the baseline visit (i.e between V1 and V2)
* Patients must have been treated with at least 2 different AEDs within the last 2 years prior to the screening visit
* The patient is capable and would like to respect all protocol requirements, include to be available for the doctor's calls and doctor's appointments at any time, follow through all protocol procedures
* The patient agrees to self - report each seizure he has experienced between 2 visits, accurately and thoroughly, in a diary he'll be provided with

Exclusion Criteria:

* Patients suffering from non-epileptic seizures
* Patients having seizures that can't be counted due to clustering.
* History of primary generalized seizures
* History of status epilepticus within 12 months prior to the screening visit
* The patient has received not permitted concomitant medications
* The patient has a progressive structural lesion in the CNS, or a progressive encephalopathy
* The patient is pregnant (or planning to become pregnant during the study) or is a lactating woman
* The patient has used Remegal previously or participated in a clinical study within 24 weeks prior to the screening visit
* The patient has experienced of any somatic disorders or psychiatric diseases and conditions which, in the opinion of the investigator, lead to health worsening or influence on the patient ability to participate in the actual clinical study
* Vulnerable patients and individuals of majority age who are subject to legal protection or unable to express their consent
* The patient has a history of chronic alcohol consumption or drug abuse within 2 years prior to the screening visit
* The patient has a known history of a severe anaphylactic reaction or severe changes in blood tests
* ALT, AST, alkaline phosphatise, total bilirubin or serum creatinine level ≥ 2 times the upper limit of normal ranges
* Clinically important abnormalities on physical examination, vital signs, ECG or laboratory test results per-formed/obtained at the screening visit that may interfere with patient's safety, compliance, or study evaluations, ac-cording to the Investigator's opinion
* The patient has a clinically significant disease, surgical condition or recent chronic consumption of non-AED medications (within 4 weeks prior to the screening visit) that might be reasonably expected to interfere with drug absorption, distribution, metabolism, excretion
* QTc interval on the ECG performed at the screening visit above 500 ms
* Diseases or concomitant medications that may prolong QTc interval

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Seizure Frequency Reduction | 12 weeks
  The assessment of efficacy will be based on the reduction of total partial seizure frequency reported in the patient's diary during the Treatment phase.

SECONDARY OUTCOMES:
Number of Seizure's-Free Days | 12 weeks
  Number seizure's-free days during the Maintenance phase
CGI | 12 weeks
  Clinical Global Impression of change (CGI) at the end of Titration and Maintenance phases
PGI | 12 weeks
  Patients' Global Impression of change (PGI) at the end of the Titration and Maintenance phases
QOLIE | 14 weeks
  Assessment of Quality of Life Instrument in Epilepsy (QOLIE) at the Baseline Visit and at the end of Maintenance Phase

CONTACTS AND LOCATIONS:
Locations (9):
- Russia (9):
  - Region psychiatric clinic, Kemerovo
  - Moscow regional psychiatric hospital, Moscow
  - State Medical University, Novosibirsk
  - State psychiatric hospital №6, Saint Petersburg
  - State Medical University, Samara
  - Republican psychiatric dispensary, Saransk
  - State Medical Academy, Smolensk
  - Medical unit of disel equipment, Yaroslavl
  - Sverdlovsk region neuropsychiatric clinic, Yekaterinburg